CLINICAL TRIAL: NCT03740360
Title: Prospective Analysis About the Utility of Contrast Enhanced Endoscopic Ultrasound and Molecular Analysis in the Study of Pancreatic Cyst
Brief Title: Contrast Enhanced Ultrasound and Molecular Analysis in the Diagnosis of Pancreatic Cyst
Status: Completed | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Other Study IDs: RHerranz; FdelaMorena (Other: HUPrincesa); CSantander (Other: HUPrincesa); PMajano (Other: HUPrincesa)
Record Dates: First submitted 2018-10-14; First posted 2018-11-14 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cyst
Keywords: Pancreatic cystic neoplasm; Molecular analysis; Mucinous cystic neoplasm; Serous cystic neoplasm; Intraductal papillary neoplasm
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Pancreatic cyst fluid and blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the use of contrast-enhanced harmonic endoscopic ultrasound (CH-EUS) and cyst fluid molecular analysis in the differential diagnosis of pancreatic cysts and the detection of malignancy.

DETAILED DESCRIPTION:
Pancreatic cyst are a frequent finding on cross-sectional imaging on general population. They are identified in up to 3% of the abdominal computed tomographies (CT) and 20% of magnetic resonance imaging (MRI) performed for other reasons but the risk of malignancy in pancreatic cysts discovered incidentally is low, representing 1-5% of the total malignant pancreatic neoplasms.

Pancreatic cysts are a broad group of pancreatic lesions that can be divided into benign and premalignant or malignant lesions. Pseudocyst and serous cystic neoplasm (SCN) don´t have malignant potential while others like mucinous cysts are premalignant lesions. But not all mucinous neoplasms have the same risk of malignancy. According to recent publications mucinous cystic neoplasm (MCN) have a potential for malignancy of around 15%, main duct intrapapillary mucinous neoplasm (MD-IPMN) of 62% and branch duct IPMN (BD-IPMN) of 25%. The correct identification of these premalignant lesions will allow to optimize the treatment and follow-up of these patients, but in many cases it is difficult to accurately differentiate between different types of cysts and their risk of malignancy. The differentiation between lmucinous and non-mucinous cysts is suboptimal, with diagnostic accuracy for CT and MRI of 61% and 50-73% with endoscopic ultrasound (EUS). The endosonographic characteristics that have been related with malignancy are the size larger than 3 cm, the presence of a solid component, wall thickening, Wirsung dilation, abrupt change of the size of the main pancreatic duct with distal atrophy of the gland and the presence of lymphadenopathies. However, endosonographic characteristics are not sufficient as an individual predictor of malignancy.

The puncture of the cyst and fine-needle aspiration (EUS-FNA) with biochemical and cytological assessment is generally indicated to differentiate between cysts and to asses for malignancy. The determination of carcinoembryonic antigen (CEA) and amylase have low specificity for the detection of malignancy and for mucinous cyst, and the cytological assessment is highly specific but lacks of sensibility (50%). So further methods are requested for an adequate detection of premalignant and malignant cyst.

Contrast-enhanced harmonic endoscopic ultrasound uses an ultrasonographic contrast agent to visualize blood flow in fine vessels and may aid in the diagnosis of pancreatic cysts by enabling assessment of the vascularization of structures such as cyst walls, septa, or mural nodules. Furthermore it allows the correct differentiation between contrast-enhanced mural nodules, that predict for malignancy, from non-enhancing mucus clots.

The molecular analysis of cyst fluid may detect mutations that are associated with premalignant cyst and with malignancy. Kirsten rat sarcoma (KRAS) gene has been related with mucinous cyst while von Hippel-Lindau gene (VHL) is present in serous cyst.

This study evaluates the use of contrast-enhanced EUS and the molecular analysis for pancreatic cyst diagnosis and malignant detection, and if their use may modify cyst management.

ELIGIBILITY:
Inclusion Criteria:

* Indeterminate pancreatic cyst > 2cm
* Pancreatic cyst > 1cm with morphological diagnosis suspicious to be mucinous etiology
* Suitable for endoscopy

Exclusion Criteria:

* Contraindication for endoscopy
* Active anticoagulant or antiplatelet therapy
* Thrombocytopenia or coagulopathy in the absence of its correction prior to the procedure
* Abscence of informed consent
* Extrapancreatic cyst
* Known pancreatic pseudocyst

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with with an imaging diagnosing pancreatic cystic neoplasm, older than 18 years old, that come to our unit during the 18 months of the study without exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Mutations in pancreatic cystic neoplasm | Baseline
  Number and type of mutations that are present on the molecular analysis of premalignant and malignant mucinous cyst.

SECONDARY OUTCOMES:
Comparison between morphological criteria and cyst fluid analysis | Baseline
  To evaluate the correlation between morphological diagnosis made by endoscopic ultrasound and diagnosis made by cyst fluid analysis (biochemical, cytological and molecular)
Increase power diagnosis with contrast-enhanced EUS | Baseline
  Percentage of pancreatic cyst that can be correctly diagnosed with contrast-enhanced EUS compared to EUS alone
Security of EUS fine-needle aspiration | 7 days
  Number of adverse events that happen during or 7 days after de procedure
Relation between pancreatic fluid and serum molecular analysis | Baseline
  Percentage of mutations that are present in both pancreatic cyst fluid and serum or only in cyst fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de la Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No